CLINICAL TRIAL: NCT04233918
Title: A Three-Part, Single-Arm, Open-Label Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Evinacumab in Pediatric Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Evaluate the Efficacy and Safety of Evinacumab in Pediatric Patients With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1500-CL-17100; 2019-001931-30 (EudraCT Number)
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: HoFH
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — evinacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Evinacumab (Experimental): Part A: Single intravenous (IV) dose Part B: IV dose every 4 weeks (Q4W) until week 20 Part C: IV dose Q4W
  Interventions: Drug: Evinacumab

INTERVENTIONS:
Drug: Evinacumab — Part A: Single IV dose Part B & C: IV dose Q4W
  Other Names: REGN1500; Evkeeza™

SUMMARY:
The primary objective for Part A of the study is to assess the pharmacokinetics (PK) of evinacumab in pediatric patients with homozygous familial hypercholesterolemia (HoFH).

The primary objective for Part B of the study is to demonstrate a reduction of low-density lipoprotein cholesterol (LDL-C) by evinacumab in pediatric (5 to 11 years of age) patients with HoFH.

The secondary objective for Part A of the study is to evaluate the safety and tolerability of evinacumab administered intravenous (IV) in pediatric patients with HoFH.

The secondary objectives for Part B of the study are:

* To evaluate the effect of evinacumab on other lipid parameters (ie, apolipoprotein B (Apo B), non-high-density lipoprotein cholesterol (non-HDL-C), total cholesterol (TC), lipoprotein a [Lp(a)]) in pediatric patients with HoFH
* To evaluate the safety and tolerability of evinacumab administered IV in pediatric patients with HoFH
* To assess the PK of evinacumab in pediatric patients with HoFH
* To assess the immunogenicity of evinacumab in pediatric patients with HoFH over time
* To evaluate patient efficacy by mutation status

DETAILED DESCRIPTION:
Part A is Phase 1b Part B is Phase 3

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of functional HoFH by either genetic or clinical criteria as defined in the protocol
2. LDL-C >130 mg/dL at the screening visit
3. Body weight ≥15 kg
4. Receiving stable maximally tolerated therapy*at the screening visit *Maximally tolerated therapy could include a daily statin.
5. Willing and able to comply with clinic visits and study-related procedures
6. Parent(s) or legal guardian(s) must provide the signed informed consent form (ICF). Patients ≥5 years of age (or above age determined by the IRB/EC and in accordance with the local regulations and requirements) must also provide informed assent forms (IAFs) to enroll in the study, and sign and date a separate IAF or ICF signed by the parent(s)/legal guardian(s) (as appropriate based on local regulations and requirements)

Key Exclusion Criteria:

1. Background pharmacologic LMT, nutraceuticals or over-the-counter (OTC) therapies known to affect lipids, at a dose/regimen that has not been stable for at least 4 weeks (8 weeks for PCSK9 inhibitors) before the screening visit and patient is unwilling to enter the run-in period
2. For patients entering Part A, unable to temporarily discontinue apheresis from the baseline visit through the week 4 visit
3. Receiving lipid apheresis, a setting (if applicable) and schedule that has not been stable for approximately 8 weeks before the screening visit or an apheresis schedule that is not anticipated to be stable over the duration of the treatment period (48 weeks).
4. Plasmapheresis within 8 weeks of the screening visit, or plans to undergo plasmapheresis during Part A or Part B
5. Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins
6. Newly diagnosed (within 3 months prior to randomization visit) diabetes mellitus or poorly controlled diabetes as defined in the protocol

Note: Other protocol-defined criteria apply

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (11):
- United States (6):
  - Regeneron Research Site, Wilmington, Delaware
  - Regeneron Research Site, Boca Raton, Florida
  - Regeneron Research Site, Kansas City, Kansas
  - Regeneron Research Center, Boston, Massachusetts
  - Regeneron Research Center, Philadelphia, Pennsylvania
  - Regeneron Research Center, Salt Lake City, Utah
- Regeneron Research Center, Westmead, New South Wales, Australia
- Regeneron Research Site, Vienna, Austria
- Regeneron Research Site, Amsterdam, Netherlands
- Regeneron Research Center, Taipei, Taiwan
- Regeneron Research Site, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Wiegman A, Greber-Platzer S, Ali S, Reijman MD, Brinton EA, Charng MJ, Srinivasan S, Baker-Smith C, Baum S, Brothers JA, Hartz J, Moriarty PM, Mendell J, Bihorel S, Banerjee P, George RT, Hirshberg B, Pordy R. Evinacumab for Pediatric Patients With Homozygous Familial Hypercholesterolemia. Circulation. 2024 Jan 30;149(5):343-353. doi: 10.1161/CIRCULATIONAHA.123.065529. Epub 2023 Oct 20. PMID 37860863

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 23 participants were screened to Part A and Part B. 6 participants were enrolled in Part A, 14 participants in Part B. 3 participants were considered screen failures. 2 withdrew consent, 1 due to Other. Participants who enrolled in Part A of study were not eligible to participate in Part B. All 20 participants completed part C.
Groups:
- Part A: Evinacumab 15mg/Kg IV: In Part A, Participants received single IV infusion of evinacumab at a dose of 15 mg/kg on Day 1.
- Part B: Evinacumab 15mg/Kg IV Q4W: In Part B, Participants received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from Day 1 up to Week 24.
- Part A to C: All participants who completed Part A received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from Day 1 up to Week 48 in Part C.
- Part B to C: All participants who completed Part B received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from Day 1 up to Week 48 in Part C.
Period: Period 1: Part A and B
Arm/Group | Part A: Evinacumab 15mg/Kg IV | Part B: Evinacumab 15mg/Kg IV Q4W | Part A to C | Part B to C
Started | 6 | 14 | 0 | 0
Completed | 6 | 14 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part C (Extension Period)
Arm/Group | Part A: Evinacumab 15mg/Kg IV | Part B: Evinacumab 15mg/Kg IV Q4W | Part A to C | Part B to C
Started | 0 | 0 | 6 | 14
Completed | 0 | 0 | 6 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: Evinacumab 15mg/Kg IV: Participants received single intravenous (IV) infusion of evinacumab at a dose of 15 milligrams per kilogram (mg/kg) on Day 1 in Part A.
- Part B: Evinacumab 15mg/Kg IV Q4W: Participants received IV infusion of evinacumab at a dose of 15 mg/kg every four weeks (Q4W) from Day 1 up to Week 24 in Part B.
- Total: Total of all reporting groups
Arm/Group | Part A: Evinacumab 15mg/Kg IV | Part B: Evinacumab 15mg/Kg IV Q4W | Total
Number analyzed (Participants) | 6 | 14 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (1.72) | 9.1 (1.94) | 9 (1.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 13 | 18
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Observed Serum Concentration (Cmax) of Evinacumab
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: At day 12
Population: Pharmacokinetic (PK) Analysis Set included all participants who received any study drug and who had at least 1 non-missing result for concentration of evinacumab following the first dose of study drug.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Part A: Evinacumab 15mg/Kg IV
Number analyzed (Participants) | 6
Milligrams per Liter (mg/L) | 238 (90.8)

2. Primary Outcome: Part A: Area Under the Serum Concentration-Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUClast) of Evinacumab
Description: AUClast was defined as area under the serum concentration time-curve from zero to the last measured concentration.
Time Frame: Up to Week 12
Population: PK Analysis Set included all participants who received any study drug and who had at least 1 non-missing result for concentration of evinacumab following the first dose of study drug.
Measure: Mean (Standard Deviation); unit: Days*Milligrams per Liter (day*mg/L)
Arm/Group | Part A: Evinacumab 15mg/Kg IV
Number analyzed (Participants) | 6
Days*Milligrams per Liter (day*mg/L) | 4576 (1568)

3. Primary Outcome: Part A: Terminal Half-Life (t1/2) of Evinacumab
Description: T1/2 was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: Up to week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Part A: Evinacumab 15mg/Kg IV
Number analyzed (Participants) | 6
Days | 7.69 [6.18 to 12.4]

4. Primary Outcome: Part B: Percent Change in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 24
Description: Percent change was calculated as 100 multiplied by (calculated LDL-C value at Week 24 minus calculated LDL-C value at baseline) divided by calculated LDL-C value at baseline.
Time Frame: Baseline to Week 24
Population: The intent-to-treat (ITT) population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Percentage of Change | -48.3 [-68.8 to -27.8]

5. Secondary Outcome: Part A and Part B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAE was defined as AE starting/worsening after first intake of study drug. TEAE included participants with both serious and non-serious AEs.
  1 participant experienced an AE during part B that was recorded after Part B database lock. This was not reflected in the reported endpoint number of participants of 10.
Time Frame: Part A: up to Week 24; Part B: up to Week 48
Population: The safety analysis set (SAF) includes all patients in Part A or Part B who received at least 1 dose or part of a dose of study drug in the respective study treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Evinacumab 15mg/Kg IV | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 6 | 14
Participants | 5 | 10

6. Secondary Outcome: Part B: Percent Change in Apolipoprotein B (Apo B) From Baseline to Week 24
Description: Percent change in Apo B from baseline to Week 24 was reported.
Time Frame: Baseline to Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Percentage of Change | -41.3 [-58.9 to -23.8]

7. Secondary Outcome: Part B: Percent Change in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 24
Description: Percent change in Non-HDL-C from baseline to Week 24 was reported.
Time Frame: Baseline to Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Percentage of Change | -48.9 [-68.1 to -29.7]

8. Secondary Outcome: Part B: Percent Change in Total Cholesterol (TC) From Baseline to Week 24
Description: Percent change in TC from baseline to Week 24 was reported.
Time Frame: Baseline to Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Percentage of Change | -49.1 [-64.9 to -33.2]

9. Secondary Outcome: Part B: Percentage of Participants With ≥50 Percent (%) Reduction in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24
Description: Percentage of participants who achieved reduction in calculated LDL-C ≥ 50% at Week 24 was reported.
Time Frame: Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Percentage of Participants | 78.6

10. Secondary Outcome: Part B: Percent Change in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 24 in Participants Who Have Negative/Negative and Null/Null Mutations
Description: Participants with HoFH was classified based on the phenotype of the Low-density lipoprotein receptor (LDLR) mutation(s), ranging from defective mutations (where the LDLR retains some LDL-binding functionality) to null or negative mutations where no functioning LDLR was expressed. Participants who have LDLR activity <15% are considered null and participants whose LDLR activity was impaired but >15% are LDLR defective. Percent change in calculated LDL-C from baseline to Week 24 in participants who have negative/negative and null/null mutations was reported.
Time Frame: Baseline to Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specified category.
Measure: Mean (Standard Error); unit: Percentage of Change
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 4
Percentage of Change
  Negative/negative mutations: number analyzed (Participants) | 3
  Negative/negative mutations | -67.7 (6.5)
  Null/Null mutations: number analyzed (Participants) | 1
  Null/Null mutations | -57.2

11. Secondary Outcome: Part B: Percent Change in Lipoprotein A (Lp[a]) From Baseline to Week 24
Description: Percent change in Lp(a) from baseline to Week 24 was reported.
Time Frame: Baseline to Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Percentage of Change | -37.3 [-42.2 to -32.3]

12. Secondary Outcome: Part B: Absolute Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline at Week 24
Description: Absolute change in LDL-C from baseline at Week 24 was reported
Time Frame: Baseline, Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Mean (Standard Error); unit: Milligrams per Deciliter (mg/dL)
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Milligrams per Deciliter (mg/dL) | -131.9 (30.0)

13. Secondary Outcome: Part B: Serum Concentration of Total Evinacumab
Description: Serum concentration of total evinacumab was reported. Pre-dose samples at week 0 were assayed and the reported value is based on actual measurement.
Time Frame: Pre-dose at Weeks 0, 4, 8, 12; End of infusion at Weeks 0.006, 4.006, 8.006, 12.006 and 24
Population: PK Analysis Set included all participants who received any study drug and who had at least 1 non-missing result for concentration of evinacumab following the first dose of study drug. Here, "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Milligrams per Liter (mg/L)
  Week 0 | 0 (0)
  Week 0.006: number analyzed (Participants) | 13
  Week 0.006 | 256 (58.0)
  Week 4 | 62.6 (22.6)
  Week 4.006 | 293 (92.3)
  Week 8 | 98.8 (37.7)
  Week 8.006 | 356 (76)
  Week 12 | 120 (46.5)
  Week 12.006 | 363 (82.1)
  Week 24: number analyzed (Participants) | 3
  Week 24 | 140 (92.5)

14. Secondary Outcome: Part B: Maximum Serum Concentration at Steady State (Cmax,ss) of Evinacumab
Description: Maximum serum concentration (Cmax,ss) steady state following drug administration.
Time Frame: Post-dose up to day 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Milligrams per Liter (mg/L) | 428.9 (113.7)

15. Secondary Outcome: Part B: Area Under the Serum Concentration-time Curve at Steady State (AUCtau.ss) of Evinacumab
Description: AUCtau.ss was defined as area under the serum concentration-time curve at steady state of evinacumab
Time Frame: Post-dose up to day 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Day*Milligrams per Liter (Day*mg/L)
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Day*Milligrams per Liter (Day*mg/L) | 7019 (2561)

16. Secondary Outcome: Part B: Minimum Serum Concentration at Steady State (Ctrough.ss) of Evinacumab
Description: Ctrough.ss was defined as minimum serum concentration at steady state of evinacumab
Time Frame: Post-dose up to day 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Milligrams per Liter (mg/L) | 171.8 (79.5)

17. Secondary Outcome: Part B: Percent Change in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 24 in Participants Who Have by Null/Null vs. Non-null/Null and Negative/Negative vs.Non-negative/Negative Mutations
Time Frame: Baseline to Week 24
Population: ITT population included all participants who received at least 1 dose or part of a dose of study drug in Part B.
Measure: Mean (Standard Error); unit: Percentage of Change
Arm/Group | Part B: Evinacumab 15mg/Kg IV Q4W
Number analyzed (Participants) | 14
Percentage of Change
  Negative/Negative: number analyzed (Participants) | 3
  Negative/Negative | -67.7 (6.5)
  Non-Negative/Negative: number analyzed (Participants) | 11
  Non-Negative/Negative | -43.0 (12.8)
  Null/Null: number analyzed (Participants) | 1
  Null/Null | -57.2 (NA) — Standard Error cannot be calculated with only 1 participant
  Non-Null/Null: number analyzed (Participants) | 13
  Non-Null/Null | -47.6 (11.3)

ADVERSE EVENTS:
Time Frame: From first dose up to week 96 (24 weeks in Part A/B + 48 weeks of treatment in Part C + 24 weeks of follow-up)
Description: Part A - up to week 24
  Part B - up to Week 48 or up to the day before the first dose in Part C for participants entering Part C; 1 participant experienced an AE during part B that was recorded after Part B database lock.
  Part C - up to a 48-week treatment period and 24-week follow-up
Groups:
- Part A Evinacumab 15mg: Participants received single intravenous (IV) infusion of evinacumab at a dose of 15 milligrams per kilogram (mg/kg) on Day 1 in Part A.
- Part B Evinacumab 15mg: Participants received IV infusion of evinacumab at a dose of 15 mg/kg every four weeks (Q4W) from Day 1 up to Week 24 in Part B.
- Part A-C Evinacumab 15mg: All participants who completed Part A received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from Day 1 up to Week 48 in Part C.
- Part B-C Evinacumab 15mg: All participants who completed Part B received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from Day 1 up to Week 48 in Part C.
Arm/Group | Part A Evinacumab 15mg | Part B Evinacumab 15mg | Part A-C Evinacumab 15mg | Part B-C Evinacumab 15mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/14 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/14 | 0/6 | 1/14
Other Adverse Events (participants affected / at risk) | 5/6 | 11/14 | 6/6 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Evinacumab 15mg (N=6) | Part B Evinacumab 15mg (N=14) | Part A-C Evinacumab 15mg (N=6) | Part B-C Evinacumab 15mg (N=14)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Evinacumab 15mg (N=6) | Part B Evinacumab 15mg (N=14) | Part A-C Evinacumab 15mg (N=6) | Part B-C Evinacumab 15mg (N=14)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 10 (10)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1) | 4 (7)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (2) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 2 (2) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (5)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poikilocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal thickening (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apheresis related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoprotein (a) increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burn oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04233918/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT04233918/SAP_001.pdf